CLINICAL TRIAL: NCT02974231
Title: Intensity-modulated Radiation Therapy From 70Gy to 80Gy in Localized Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Other Study IDs: ICL_2014_0002
Record Dates: First submitted 2016-10-10; First posted 2016-11-28 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

INTERVENTIONS:
Radiation: Intensity-modulated radiation therapy

SUMMARY:
The objective is to report outcomes,including grade ≥2 overall late rectal and urinary toxicity and biochemical control rates in patients treated with IMRT (70 gy, 74 Gy and 80 Gy)

ELIGIBILITY:
Inclusion Criteria:

Consecutive patients from June 2000 to December 2010 with

* untreated histologically confirmed adenocarcinoma of the prostate
* stage T1c-T4 N0 M0 according to the 1992 American Joint Committee on Cancer staging system

Exclusion Criteria:

* Patients with positive pelvic lymphadenectomy or radiological positives nodes

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients records would be extracted from the electronic health record system of Institut de Cancérologie de Lorraine
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2014-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
grade≥ 2 overall late rectal 5 years after the end of radiotherapy | 60 months